CLINICAL TRIAL: NCT00924417
Title: A Distraction Protocol for Peripheral IV Placement in the Pediatric Emergency Department
Brief Title: A Distraction Protocol for Peripheral Intravenous (IV) Placement in the Pediatric Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Fellow unable to complete enrollment before completing training.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Elizabeth C. Powell, Professor of Pediatrics, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMRCIRB#2008-13630
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Pain
Keywords: Pain associated with peripheral intravenous line placement
MeSH Terms: conditions — Pain | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Distraction (Experimental): Parent given brief teaching session on concept of distraction, and parent and child given 3 "distraction" toys/tools to assist with peripheral intravenous line placement.
  Interventions: Behavioral: Distraction
- Routine care (Other): Patient managed as routine care.
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Routine Care — Parent given placebo intervention that entails brief information about what is routine care for intravenous line placement in the emergency department
  Arms: Routine care
Behavioral: Distraction — Parent given brief information about the cognitive behavioral technique known as distraction. Parent and child then given 3 distraction "toys/tools" to assist with peripheral intravenous line placement.
  Arms: Distraction

SUMMARY:
This is a randomized, controlled trial of a distraction protocol for peripheral intravenous line placement in the pediatric emergency department. Patients and parents will be randomized to one of two interventions: routine care or a teaching session about the cognitive technique known as distraction. The study seeks to enroll children ages 4-9, who are cognitively normal, who are without significant chronic medical illness, who are receiving intravenous line placement as part of routine care in the pediatric emergency department. Study investigators hypothesize that patients in the intervention group will report less pain than patients in the control group.

DETAILED DESCRIPTION:
Routine care patients will have intravenous lines placed in the usual manner.

Intervention patient families will have a teaching session about distraction techniques, and distraction will be used during the intravenous line placement.

ELIGIBILITY:
Inclusion Criteria:

* Ages 4 - 9
* Requiring IV placement for medical care in emergency department
* Child cognitively normal

Exclusion Criteria:

* No significant chronic medical conditions
* No IV in past 3 years

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Faces Pain Scale Revised as reported by child | To be completed 5 minutes after IV placement

SECONDARY OUTCOMES:
Visual Analog Scales to be completed by parent in order to measure: parent distress, patient/child pain, patient/child distress | 5 minutes after IV completion

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Powell, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States